CLINICAL TRIAL: NCT04930354
Title: A Phase 1 Open-Label, Multiple Dose, Two Part Dose Escalation Study of ECP-1014 as a Treatment for Patients With Solid Tumor Cancers
Brief Title: ECP-1014 Treatment for Patients With Solid Tumor Cancers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Euclises Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECP-1014-001
Record Dates: First submitted 2021-05-26; First posted 2021-06-18 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Solid Tumor

STUDY DESIGN:
Intervention Model Description: Sequential study model; first dose is 10mg, then 20mg, 40mg, 80mg and 160mg.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Single arm dose escalation study; ECP1014 oral capsule of10mg, 20mg, 40mg, 80mg and 160mg given once daily for 28 days
  Interventions: Drug: ECP-1014

INTERVENTIONS:
Drug: ECP-1014 — Patients will be selected who (1) have failed all standard of care therapy (relapsed/refractory) or (2) have relapsed and are not a candidate for an available standard of care therapy as assessed by the investigator (such as, but not limited to, colorectal cancer (CRC), Non-Small Cell Lung Cancer (NSCLC), head and neck, etc.) with COX-2 overexpression, ultimately resulting in elevated production of prostaglandin E2 (PGE2).
  Other Names: GIBH-1014

SUMMARY:
The primary objective of this study is to evaluate the safety, tolerability, pharmacokinetics, and optimal recommended Phase 2 dose (RP2D) during a 28-day dosing period of ECP-1014 in patients with solid tumors and by evaluation of dose limiting toxicities.

DETAILED DESCRIPTION:
This is a single arm, single-center, open-label, ascending dose study in which dose escalation will be determined based on safety and tolerability. Up to a total of 6 cohorts of patients will be enrolled unless additional intermediate doses are studied, not to exceed the maximal dose per protocol.

There are 2 Parts to this study.

* Part 1 involves enrolling sequential cohorts of patients into a dose-escalation design, in which doses are assessed for safety/tolerability.
* Part 2 involves randomizing a cohort of patients to the highest and second-highest tolerated doses as identified in Part 1.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is male or female 18 years of age or older
2. The patient or legal representative has voluntarily signed and dated an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written informed consent.
3. Female patients must be of non-childbearing potential (surgically sterile or post-menopausal for at least 1 year) or be practicing a highly effective contraception method from consent to at least 30 days after the last dose of study medication. Highly effective contraception methods include: vasectomized partner (at least 6 months prior to dosing); double barrier (diaphragm with spermicide; condoms with spermicide); intrauterine device; implanted or intrauterine hormonal contraceptives in use for at least 6 consecutive months prior to study dosing and throughout the study duration; oral, patch, or injected contraceptives in use for at least 3 consecutive months prior to study dosing.
4. Male patients will be required to practice highly effective contraception methods such as: having had a vasectomy, double barrier (condoms with spermicide) or abstinence.
5. Female patients of childbearing potential have a negative pregnancy test (serum β human chorionic gonadotropin [HCG]) during screening and ≤ 24 hours prior to dosing and are not lactating.
6. Histologically confirmed solid malignant tumors, which are suspected to over express COX-2 by elevations in urinary PGE-M, such as, but not limited to colorectal, non-small cell lung cancer, head and neck, etc.
7. Patients who (1) have failed all standard of care therapy (relapsed/refractory) or (2) have relapsed and are not a candidate for an available standard of care therapy as assessed by the investigator.
8. Elevated urinary PGE-M levels at least 1.5 times the upper normal limits (Males 10.4+1.5, Females 6.0+0.7 ng/mg creatinine).
9. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2 and able to comply with protocol.
10. Patients with treated brain metastases are eligible if there is no evidence of progression for at least 2 weeks after CNS-directed treatment, as ascertained by clinical examination and brain imaging during the screening period.
11. Life Expectancy ≥ 12 weeks.
12. Normal organ function as defined below:

    1. platelets ≥100,000/mcL
    2. total bilirubin ≤1.5X the institutional upper limit of normal (ULN)
    3. AST(SGOT)/ALT(SGPT) <2.5X institutional ULN or <5X institutional ULN in the presence of liver metastases
    4. creatinine clearance ≥45 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal (use Cockcroft-Gault formula)
    5. absolute neutrophil count ≥1,500/mcL.
13. No prior history of myocardial infarction, angina pectoris, coronary artery bypass graft (CABG) within 6 months prior to starting study treatment
14. No congestive heart failure, clinically significant cardiac arrhythmias, complete left bundle branch block, high-grade AV block, left ventricular ejection fraction <50% evaluated by ECHO or MUGA requiring treatment.
15. No increased QTCF (>450 for men and >470 for women).
16. No NSAIDS, full dose oral anticoagulation such as warfarin within 2 weeks of screening.
17. No gastric acid-reducing agents.
18. Avoid strong inhibitors or inducers of CYP450
19. The patient is willing and able to understand the study procedures and to comply with the study protocol.

Exclusion Criteria:

1. Receiving other investigational drugs or participated in a clinical investigation trial of an agent within 30-days prior to or washout of at least 5 half-lives of the investigational drug prior to Day 1 (dosing of ECP-1014), whichever is longest.
2. Patients with known hypersensitivity to COX-2, aspirin, or other NSAIDs, history of asthma, urticaria, or allergic-type reactions after taking aspirin or other NSAIDs. And those with history of allergic-type reactions to sulfonamides.
3. Significant gastrointestinal abnormalities that may affect absorption (e.g., gastric bypass, short gut syndrome).
4. History of gastric ulcer or gastrointestinal bleed.
5. Known human immunodeficiency virus (HIV), acute or chronic hepatitis B virus surface antigen or (HBsAg) hepatitis C virus (HCV).
6. Ongoing ≥ CTCAE grade 2 toxicity (except alopecia) due to prior cancer therapy.
7. Patient has a condition that precludes ability to consume study medication.
8. Concomitant disease or condition that, in the clinical judgment of the treating physician, is likely to prevent the subject from complying with any aspect of the protocol or that may put the subject at unacceptable risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
This is a safety and tolerability-based study in which the MTD may be determined | 28 days
  All AEs will be classified with respect to the MedDRA System Organ Class (SOC) and preferred term. The number and percent of patients who report treatment-emergent adverse events (TEAEs) will be summarized for each treatment group. Additional summaries by severity, relationship, and subgroup will be presented. Serious AEs (SAEs) will be summarized similarly. Clinical chemistry, hematology, and urinalysis will be preformed and changes will be compared to baseline.

SECONDARY OUTCOMES:
Plasma for Peak Plasma Concentration (Cmax) | Day 1 at Hours 0 (immediately pre-morning dose), and Hours 0.5, 1.0, 2, 3, 4, 6, 8, 10, 12, 18 and 24. The patient will return to the clinic on the morning of Day 5 after fasting
  A 24-hour intensive blood plasma sampling for pharmacokinetic concentration determination will be performed on Day 1 at Hours 0 (immediately pre-morning dose), and Hours 0.5, 1.0, 2, 3, 4, 6, 8, 10, 12, 18 and 24. Patients will be required to remain in-clinic overnight for this sampling.
  The patient will return to the clinic on the morning of Day 5 after fasting from the evening before. Following the Hour 0 (trough) PK sample, the subject will be given their morning dose of study medication. Additional PK samples will be collected at Hours 0.5, 1.0, 2, 3, 4, 6, 8, 10, 12, 18 and 24.
Urine for PGE-M levels | Pretreatment, Days 5 & 28
  Exploratory biomarkers such as urinary PGE-M will be measured to assess the pharmacodynamic effects of the investigational drug. Starting the morning of Day 4 through the morning of Day 5, a 24-hour urine collection will be performed to allow for assessment of ECP-1014 and metabolite excretion.
Plasma for Area Under the Curve (AUC) | Day 1 at Hours 0 (immediately pre-morning dose), and Hours 0.5, 1.0, 2, 3, 4, 6, 8, 10, 12, 18 and 24. The patient will return to the clinic on the morning of Day 5 after fasting
  A 24-hour intensive blood plasma sampling for pharmacokinetic concentration determination will be performed on Day 1 at Hours 0 (immediately pre-morning dose), and Hours 0.5, 1.0, 2, 3, 4, 6, 8, 10, 12, 18 and 24. Patients will be required to remain in-clinic overnight for this sampling.
  The patient will return to the clinic on the morning of Day 5 after fasting from the evening before. Following the Hour 0 (trough) PK sample, the subject will be given their morning dose of study medication. Additional PK samples will be collected at Hours 0.5, 1.0, 2, 3, 4, 6, 8, 10, 12, 18 and 24.
Plasma for Half-life (t1/2) | Day 1 at Hours 0 (immediately pre-morning dose), and Hours 0.5, 1.0, 2, 3, 4, 6, 8, 10, 12, 18 and 24. The patient will return to the clinic on the morning of Day 5 after fasting
  A 24-hour intensive blood plasma sampling for pharmacokinetic concentration determination will be performed on Day 1 at Hours 0 (immediately pre-morning dose), and Hours 0.5, 1.0, 2, 3, 4, 6, 8, 10, 12, 18 and 24. Patients will be required to remain in-clinic overnight for this sampling.
  The patient will return to the clinic on the morning of Day 5 after fasting from the evening before. Following the Hour 0 (trough) PK sample, the subject will be given their morning dose of study medication. Additional PK samples will be collected at Hours 0.5, 1.0, 2, 3, 4, 6, 8, 10, 12, 18 and 24.
Plasma for Time to Maximum Plasma Concentration (Tmax) | Day 1 at Hours 0 (immediately pre-morning dose), and Hours 0.5, 1.0, 2, 3, 4, 6, 8, 10, 12, 18 and 24. The patient will return to the clinic on the morning of Day 5 after fasting
  A 24-hour intensive blood plasma sampling for pharmacokinetic concentration determination will be performed on Day 1 at Hours 0 (immediately pre-morning dose), and Hours 0.5, 1.0, 2, 3, 4, 6, 8, 10, 12, 18 and 24. Patients will be required to remain in-clinic overnight for this sampling.
  The patient will return to the clinic on the morning of Day 5 after fasting from the evening before. Following the Hour 0 (trough) PK sample, the subject will be given their morning dose of study medication. Additional PK samples will be collected at Hours 0.5, 1.0, 2, 3, 4, 6, 8, 10, 12, 18 and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, MD, Principal Investigator — The Sixth Affiliated Hospital Sun Yat-sen University, Guangzhou, China
Locations (1):
- The Sixth Affiliated Hospital Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No